CLINICAL TRIAL: NCT07139730
Title: Effect of Nebulized Lignocaine on the Stress Response of Endotracheal Intubation in Pediatrics Undergoing Tonsillectomy Operation ; A Randomized Controlled Clinical Trial
Brief Title: Effect of Nebulized Lignocaine on the Stress Response of Endotracheal Intubation in Pediatrics Undergoing Tonsillectomy Operation Monitored by Rise in Serum Cortisol Level Post Intubation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Sayed Frag Ahmed, doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: stress Response of ETT
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Stress Response
MeSH Terms: conditions — Fractures, Stress | interventions — Lidocaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Effect of Nebulized Lignocaine on the stress Response of Endotracheal Intubation in pediatrics unde (Experimental)
  Interventions: Drug: Lignocaine 2% concentration solution

INTERVENTIONS:
Drug: Lignocaine 2% concentration solution — the effect of preoperative nebulized lidocaine on the stress response to intubation, monitored by rise in serum cortisol level post intubation

SUMMARY:
This randomized clinical trial aims to is examining the effect of preoperative nebulized lidocaine on the stress response to intubation, monitored by rise in serum cortisol level post intubation

DETAILED DESCRIPTION:
Endotracheal intubation is a routine and often critical procedure performed in patients who require airway management, particularly during surgeries, emergency interventions, or in cases of respiratory failure. While essential, the process of intubation can provoke significant hemodynamic changes in patients, including fluctuations in heart rate, blood pressure, and other vital parameters. These hemodynamic responses are primarily a result of the stimulation caused by the mechanical manipulation of the airway and the associated stress response. (1,2).

The stress response to intubation is mainly mediated by the sympathetic nervous system, leading to an increase in catecholamine release, which in turn causes an elevation in heart rate and blood pressure. In certain vulnerable populations, such as those with pre-existing cardiovascular conditions, these changes can be problematic and increase the risk of complications such as arrhythmias, myocardial ischemia, and cerebrovascular events. (2, 3).

Lignocaine is a local anesthetic that has been shown to have antiarrhythmic properties and can be administered through various routes to reduce the stress response associated with endotracheal intubation. It can be delivered intravenously or via inhalation through a nebulizer. The intravenous route (IV) is commonly used in clinical practice to provide systemic analgesia and reduce sympathetic stimulation. Nebulized lignocaine, on the other hand, delivers the drug directly to the airway and has been proposed as a potential alternative for reducing the hemodynamic impact of intubation while also minimizing systemic side effects. (4,5,6).

Previous studies have suggested that both intravenous and nebulized lignocaine may be effective in attenuating the hemodynamic response to intubation. However, there remains a gap in understanding regarding the comparative efficacy, optimal dosing, and side-effect profiles of these two administration methods. While both approaches have been used in various clinical settings, there has been limited research examining their direct effects and comparison in a controlled, randomized trial setting. (7) .

ELIGIBILITY:
Inclusion Criteria: 1. Elective tonsillectomy operation 2- pediaterics below 9 years old 3- ASA I OR II

-

Exclusion Criteria: 1- emergency cases as bleeding tonsills 2- ASA III OR IV

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
effect on serum cortisol level 2 minutes after intubation | baseline
effect on serum cortisol level 2 minutes after intubation | baseline
  effect on serum cortisol level 2 minutes after intubation to asses decrease in stress response